CLINICAL TRIAL: NCT05651802
Title: Prophylactic Cranial Irradiation and Brain MRI Follow-up Versus Brain MRI Follow-up Alone in Patients With Limited-stage Small Cell Lung Cancer Who Achieved Complete Remission After Definitive Radio-chemotherapy: a Prospective Randomized Trial
Brief Title: PCI and Brain MRI Follow-up vs Brain MRI Follow-up Alone in Limited-stage SCLC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Sun Yat-sen University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hu Xiao, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCI+MRI vs. MRI
Record Dates: First submitted 2022-12-02; First posted 2022-12-15 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Small Cell Lung Cancer Limited Stage
Keywords: prophylactic cranial irradiation; brain MRI follow-up; prognosis
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Patients who are randomized to control arm are those who have achieved complete remission of tumor after definitive radio-chemotherapy and will receive PCI and regular brain MRI follow-up.
  Interventions: Radiation: Prophylactic cranial irradiation; Radiation: Thoracic radiotherapy; Drug: Chemotherapy
- Study arm (Experimental): Patients who are randomized to study arm are those who have achieved complete remission of tumor after definitive radio-chemotherapy and will receive regular brain MRI follow-up alone.
  Interventions: Radiation: Thoracic radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Prophylactic cranial irradiation — Prophylactic cranial irradiation (PCI) is actually a habitual statement. It is a technique used to eliminate tiny metastatic lesions that have already existed in the brain, but can not be found by brain MRI and other inspection methods.
  Arms: Control arm
Radiation: Thoracic radiotherapy — Thoracic radiotherapy is a local treatment of tumors located in the chest using ionizing radiation.
Drug: Chemotherapy — Chemotherapy is the abbreviation of chemical drug therapy. It is a treatment method that uses chemical drugs to prevent the proliferation, invasion and metastasis of cancer cells, and finally kill cancer cells.

SUMMARY:
At present, prophylactic cranial irradiation (PCI) is part of standard care for patients with limited-stage small cell lung cancer (SCLC) who have achieved good response after definitive thoracic radiotherapy and chemotherapy. However, the value of PCI is being challenged in the era when MRI examination of brain has been popularized.

The goal of this clinical study is to compare PCI and regular brain MRI follow-up (control arm) and regular brain MRI follow-up alone (study arm) in patients with limited-stage SCLC who have received definitive radiotherapy and chemotherapy and acheived complete remission (CR) of tumor.

The main questions to answer are:

1. Whether the 2-year brain metastasis-free survival rate of the study group is not inferior to that of the control group.
2. The difference of 2-year overall survival rate between the control group and the study group.
3. Whether the patients in the study group have better overall quality of life than those in the control group.

Participants will randomly receive either PCI and regular brain MRI follow-up or regular brain MRI follow-up alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven diagnosis of SCLC.
* Age ≥ 18 years.
* Karnofsky performance status ( KPS) ≥80.
* The limited-stage is defined as the tumor confined to one side of the chest, including ipsilateral hilar, bilateral mediastinum, and bilateral supraclavicular lymph nodes. (The definition of metastatic lymph nodes is that the short diameter ≥ 1cm or PET-CT shows increased metabolism with SUV≥2.5, or proved by mediastinoscopy/EBUS/TBNA biopsy. The thickness of pleural effusion on chest CT is less than 1cm (unless cytology proves to be malignant pleural effusion). According to 8th AJCC/UICC TNM staging system, it is the I-IIIC without intrapulmonary metastasis.
* Patients who have received definitive chest radiotherapy and chemotherapy and achieved complete remission of tumor within 4-6 weeks after the end of radio-chemotherapy (in accordance with the Response Evaluation Criteria in Solid Tumors v.1.1 including enhanced CT scan of chest and abdomen, enhanced brain MRI, bone scan and tumor markers).
* Good follow-up compliance;
* Fully understand this study, and voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients with a history of malignant tumors (past or concurrent) within 5 years, excluding papillary thyroid cancer, non-malignant melanoma skin cancer and cervical carcinoma in situ.
* Patients who have received radical surgery (excluding biopsy).
* Patients with psychiatric history, pregnancy and lactation.
* Uncontrolled diabetes, hypertension, severe active infection.
* Patients with chronic diseases of central nervous system.
* Patients with contraindications of brain MRI examination.
* Other situations deemed unsuitable by the doctor in charge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
2-year brain metastasis-free survival estimated with kaplan-Meier method | Up to 2 years
  To test with a one-sided significance of 5% whether for the treatment of limited-stage SCLC patients, brain MRI follow-up alone is non-inferior in terms of 2-year brain metastasis-free survival compared to PCI and brain MRI follow-up. Participants were monitored for up to 2 years. The brain metastasis-free survival time is defined as the time between the date of the first treatment until the date of first documented diagnosis of brain metastasis or the date of death from any cause.

SECONDARY OUTCOMES:
2-year overall survival estimated with kaplan-Meier method | Up to 2 years
  To compare 2-year overall survival between patients who receive brain MRI follow-up alone and those who receive both PCI and brain MRI follow-up, with kaplan-Meier estimates. Participants were monitored for up to 2 years. The overall survival time is defined as the time between the date of the first treatment until the date of death from any cause.
Intra-cranial progressive patterns | Up to 2 years
  To compare the intra-cranial progressive patterns between patients who receive brain MRI follow-up alone and those who receive both PCI and brain MRI follow-up within 2 years. Intra-cranial progression is evaluated via the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. In this study, Intra-cranial progressive disease is defined as the new lesions developed in the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Hu, MD, PhD, Principal Investigator — Zhejiang Cancer Hospital
Locations (2):
- China (2):
  - Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No